CLINICAL TRIAL: NCT00232518
Title: Randomised Controlled Clinical Trial of the Effect of Therapeutic Hookworm Infection in Allergic Rhinoconjunctivitis
Brief Title: Randomised Controlled Clinical Trials of the Effect of Therapeutic Hookworm Infection in Allergic Rhinoconjunctivitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GR076306
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2007-05-07 (Estimated); Status verified 2005-04

CONDITIONS: Rhinitis, Allergic, Perennial; Hayfever; Allergy
Keywords: immune system; infection; allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis, Allergic, Seasonal; Hypersensitivity; Infections; Rhinitis, Allergic

INTERVENTIONS:
Procedure: Infection with hookworm larvae

SUMMARY:
There has been considerable debate over the last 30 years about the interaction between asthma and parasitic infection. It has been suggested that at least part of the reason for the increasing prevalence of asthma in the developed world is a decrease in parasite infections resulting from improved living conditions with economic development. Our previous studies in Ethiopia suggest that hookworm infection may be particularly important in this process.

To establish definitively whether parasites can protect against allergic disease, and specifically asthma, ultimately requires a randomised clinical trial of parasite infection in patients with asthma. We, the researchers at the University of Nottingham, have completed a study in normal volunteers to establish the dose of hookworms necessary to generate infection at the level shown to be protective in population surveys, and shown that infection is well tolerated. We now propose two randomised placebo-controlled double blind clinical trials. The first will test the effectiveness of hookworm infection in reducing symptoms in allergic patients with rhinitis, and will also serve to allow us to check the likely safety of hookworm infection in asthma. Assuming that the results of this study are favourable, we will then carry out a trial of hookworm infection in asthma. We will also take the opportunity during both of these studies to investigate the cellular mechanisms of the effect of hookworm infection on the immune system.

DETAILED DESCRIPTION:
Epidemiological evidence suggests that human hookworm infection is associated with a reduced risk of asthma and allergic disease. This association is potentially important not only to understanding the aetiology of asthma and allergic disease, but also because it suggests that hookworms or their products might be therapeutically effective in these conditions. To test the hypothesis that hookworms protect against asthma ultimately requires a clinical trial.

We have carried out a dose-ranging study to establish the dose of hookworm larvae necessary to generate infection at the intensity shown to be protective in epidemiological studies, with acceptable side effects, and now propose to test the effect of 12 weeks of hookworm infection at this level of intensity in two randomised placebo controlled clinical trials. The first will be in patients with allergic rhinoconjunctivitis, to determine whether hookworm infection improves rhinitis symptoms and also, because these patients will have measurable airway responsiveness, to determine whether airway responsiveness changes during the lung migration phase of the hookworm life cycle. If this study confirms that hookworm infection does not increase airway responsiveness, we will proceed to a similar trial in patients with asthma.

In both studies we will also measure a range of relevant immunological parameters to explore the relation between these parameters and expression of the allergic and asthmatic phenotypes.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of allergic rhinitis
* Measurable airway responsiveness to AMP
* Negative hookworm serology
* Positive skin prick tests to D.pteronyssinum, cat fur or grass pollen

Exclusion Criteria:

* History of asthma
* History of anaemia
* History of severe allergic reaction or anaphylaxis
* Possible or planned pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-09; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Maximum change from baseline in airway responsiveness to adenosine 5'-monophosphate (AMP) during the lung migration phase of hookworm infection.

SECONDARY OUTCOMES:
Change from baseline in rhinoconjunctivitis quality of life questionnaire score
allergen skin wheal response
mean daily peak flow
total- and specific serum IgE titres
acidic mammalian chitinase, cytokine profiles, other inflammatory markers
occurrence of adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: John Britton, Principal Investigator — University of Nottingham; David Prichard, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, United Kingdom